CLINICAL TRIAL: NCT05128838
Title: RISE (Reinvent, Integrate, Strengthen, Expand) Self-Management Program for Cancer Survivors: A Feasibility Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arash Asher, MD (Other)
Responsible Party: Sponsor-Investigator, Arash Asher, MD, Associate Professor, Medicine and Physical Medicine and Rehabilitation, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2020-28-SLEIGHT-RISE
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Survivorship
Keywords: Cancer Survivor; Self-management; Lifestyle; Survivorship
MeSH Terms: conditions — Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RISE Intervention (Experimental): Working one-on-one with the PI (a licensed occupational therapist (OT) and behavior change expert), participants will set goals and develop practical strategies in order to establish sustainable positive habits around lifestyle areas such as physical activity, nutrition, stress management, sleep, self-efficacy, and spiritual well-being. Motivational interviewing, cognitive behavioral therapy, and patient education will accompany intensive collaborative problem-solving and creation of accountability structures to create increased self-efficacy for health self-management.
  Interventions: Other: RISE (Reinvent, Integrate, Strengthen, Expand) Intervention

INTERVENTIONS:
Other: RISE (Reinvent, Integrate, Strengthen, Expand) Intervention — Working one-on-one with the PI (a licensed occupational therapist (OT) and behavior change expert), participants will set goals and develop practical strategies in order to establish sustainable positive habits around lifestyle areas such as physical activity, nutrition, stress management, sleep, self-efficacy, and spiritual well-being. Motivational interviewing, cognitive behavioral therapy, and patient education will accompany intensive collaborative problem-solving and creation of accountability structures to create increased self-efficacy for health self-management. In summary, the RISE intervention includes three components: patient education, internalization of self-determination, and habit formation.

SUMMARY:
This is a prospective feasibility study using a convenience sample of cancer survivors from Cedars-Sinai and its surrounding catchment area. As this study will be primarily focused on optimization of the RISE (Re-invent, Integrate, Strengthen, Expand) protocol, there will be no control group or randomization of participants. The RISE intervention is informed by the principles of Lifestyle Redesign, an occupational therapy-based therapeutic technique focused on measurable, individually-tailored, health-related goals. All participants will complete the 13-session RISE intervention. Sessions will occur weekly or biweekly. Measures will be completed at baseline (session #0) and post-intervention (session #12), with repeat survey measures at midpoint (session #6). There will also be a follow-up timepoint 12 weeks after the final session, at which time some measures will be completed to assess long-term maintenance of self-efficacy improvement.

ELIGIBILITY:
Inclusion Criteria:

1. History of cancer diagnosis within two years prior to enrollment
2. Completed all primary cancer treatment (surgery, radiation, and/or chemotherapy) at least 12 weeks before initial RISE session. Long-term hormonal/biologic therapy is acceptable.
3. Identified by oncologist, by medical record, or by self-report as having at least one lifestyle-related risk factor for cancer recurrence. Lifestyle-related risk factors include:

   * BMI of 25 or higher;
   * Sedentary lifestyle, defined as physical activity of less than 150 minutes per week of moderate-intensity aerobic activity OR less than 75 minutes per week of vigorous aerobic activity;
   * Non-adherence to dietary recommendations, including intake of less than five portions or servings (at least 400g or 15oz in total) of fruit/vegetables per day; consumption of ultra-processed foods more than once a week, defined as foods high in fat, starches or sugars (including "fast foods", pre-prepared dishes, bakery foods, and desserts); consumption of red/processed meats above 500g or 18oz cooked weight per week, and/or intake of more than 3 alcoholic beverages a week, per patient report;
   * Smoking cigarettes or e-cigarettes;
   * Patient self-report of high unmanaged stress, as measured by a score of 1, 2, or 3 out of 5 (responses indicating a clinically relevant level of emotional/mental stress) on at least one of two items from the PROMIS Global 10: "How often have you been bothered by emotional problems such as feeling anxious, depressed or irritable?" and "In general, how would you rate your mental health, including your mood and your ability to think?
   * Patient self-report of fatigue (either due to too little sleep, too much sleep, or any other cause), as measured by a score of 1, 2, or 3 out of 5 (responses indicating a clinically relevant level of fatigue) on a single item from the PROMIS Global 10: "How would you rate your fatigue on average?".
4. Treating and/or study physician clearance to participate in this study's program and to work toward World Cancer Research Fund and American Institute for Cancer Research (WCRF/AICR) lifestyle recommendation-related goals.
5. Age >18 years
6. Ability to read, write, and understand English.
7. Written informed consent obtained from participant and ability for participant to comply with the requirements of the study.

Exclusion Criteria:

1. Cognitive issues substantially affecting patient's ability to participate in the study, as determined by the PI or study physician.
2. Planning to have active anti-cancer treatment (including radiation, chemo, and/or major surgery) within 6 months after initial RISE session. Long-term hormonal/biologic therapy is acceptable.
3. Known metastatic disease (stage IV cancers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
RISE program feasibility will be measured by tracking participant attrition rate. RISE program will be considered feasible if ≥80% of study participants complete ≥10 RISE sessions. | Up to 38 weeks.
  All participants will complete the 13-session RISE intervention. RISE program will be considered feasible if ≥80% of study participants complete ≥10 RISE sessions of the total 13 sessions.

SECONDARY OUTCOMES:
To measure participant acceptability of the RISE program through a survey at the final RISE session. | Up to 24 weeks.
  The RISE Satisfaction Survey will use a Likert scale to ask to what extent participants found that the program improved their confidence in their ability to manage their own health, as well as how much it improved their overall well-being. Two questions are measured on a scale of 0-4, where higher scores indicate higher satisfaction rate. The remaining questions are measured on a scale of 0-10, where higher scores indicate more positive feedback and higher acceptability of the program. Participants will also have the opportunity to rate the RISE instructor (on a scale of 0-10, 10 being the best possible rating) and will include an open text box for suggestions for future iterations of the program.
To test the impact of the RISE intervention on participant self-efficacy, as measured by the PROMIS General Self-Efficacy Short Form questionnaire. | Up to 24 weeks.
  he PROMIS General Self-Efficacy Short Form questionnaire consists of 4 questions that asks the subject to rate their confidence levels in managing various situations, problems, and events. Each question is answered on a scale of 1-5, where higher scores indicate the highest level of confidence. The questionnaire responses at baseline and end of study will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Asher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No